CLINICAL TRIAL: NCT02378805
Title: European Alport Therapy Registry - European Initiative Towards Delaying Renal Failure in Alport Syndrome: Current and Novel Therapies
Brief Title: Alport Therapy Registry - European Initiative Towards Delaying Renal Failure in Alport Syndrome
Acronym: Alport-XXL
Status: Recruiting | Type: Observational
Sponsor: University Hospital Goettingen (Other)
Collaborators: Society for Pediatric Nephrology (Germany) (Other)
Responsible Party: Principal Investigator, Prof. Dr. O. Gross, Prof. Dr. Oliver Gross, University Hospital Goettingen
Other Study IDs: Alport-UMG2010
Record Dates: First submitted 2015-02-26; First posted 2015-03-04 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Alport Syndrome; Hereditary Kidney Disease; Pediatric Kidney Disease; Thin Basement Membrane Disease; Familial Benign Hematuria
Keywords: Alport syndrome; thin basement membrane disease; familial benign hematuria
MeSH Terms: conditions — Nephritis, Hereditary; Hematuria, Benign Familial | interventions — Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Spironolactone; finerenone; paricalcitol; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- no-T: untreated patients: untreated patients, typically uncles or grandfathers of present patients. No Intervention (means no therapy until CKD stage V, on renal replacement therapy)
- T-III: late therapy in patients: patients treated with medications with low eGFR (below 60 ml/min) (starts at patients with CKD stages III and IV).
  Interventions: Drug: ACE-inhibitor; Drug: Angiotensin-receptor blocker (ARB); Drug: HMG-Coenzyme inhibitor (statin); Drug: Spironolactone or Finerenone; Drug: Paricalcitol; Drug: SGLT2 inhibitor
- T-II: early therapy in patients: therapy starts in patients with albuminuria >300mg/gCreatinine and eGFR higher than 60 ml/min.
  Interventions: Drug: ACE-inhibitor; Drug: Angiotensin-receptor blocker (ARB); Drug: HMG-Coenzyme inhibitor (statin); Drug: Spironolactone or Finerenone; Drug: Paricalcitol; Drug: SGLT2 inhibitor
- T-I: very early therapy in patients: therapy starts in patients with microhematuria only (usually at birth) or microalbuminuria (30-300 mg albumin per gCreatinine).
  Interventions: Drug: ACE-inhibitor; Drug: Angiotensin-receptor blocker (ARB); Drug: HMG-Coenzyme inhibitor (statin); Drug: Spironolactone or Finerenone; Drug: Paricalcitol; Drug: SGLT2 inhibitor
- no therapy in heterozygous patients: heterozygous patients without therapy
- therapy in heterozygous patients: heterozygous patients with therapy (which also can be divided into subgroups stage T-0, I, II, III)
  Interventions: Drug: ACE-inhibitor; Drug: Angiotensin-receptor blocker (ARB); Drug: HMG-Coenzyme inhibitor (statin); Drug: Spironolactone or Finerenone; Drug: Paricalcitol; Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: ACE-inhibitor — observational study
  Groups: T-I: very early therapy in patients; T-II: early therapy in patients; T-III: late therapy in patients; therapy in heterozygous patients
Drug: Angiotensin-receptor blocker (ARB) — observational study
  Groups: T-I: very early therapy in patients; T-II: early therapy in patients; T-III: late therapy in patients; therapy in heterozygous patients
Drug: HMG-Coenzyme inhibitor (statin) — observational study
  Groups: T-I: very early therapy in patients; T-II: early therapy in patients; T-III: late therapy in patients; therapy in heterozygous patients
Drug: Spironolactone or Finerenone — observational study
  Groups: T-I: very early therapy in patients; T-II: early therapy in patients; T-III: late therapy in patients; therapy in heterozygous patients
Drug: Paricalcitol — observational study!
  Groups: T-I: very early therapy in patients; T-II: early therapy in patients; T-III: late therapy in patients; therapy in heterozygous patients
Drug: SGLT2 inhibitor — observational study
  Groups: T-I: very early therapy in patients; T-II: early therapy in patients; T-III: late therapy in patients; therapy in heterozygous patients

SUMMARY:
The hereditary type IV collagen disease Alport syndrome leads to kidney failure early in life. Currently there are no specific medications approved for treatment, however, several therapies have been evaluated preclinically and could improve outcome. For that reason, this non-interventional, observational study investigates, if medications (1) delay disease progression; (2) delay time to kidney failure; (3) improve life-expectancy compared to untreated patients (relatives). This observational study started in 2006 as an European registry. Since 2019, this registry has been expanded to "Alport XXL" via the International Alport Alliance as a global effort across all continents. From 2020 on to present, "Alport XXL" has a special focus on the outcomes of early therapy in young patients on ACE-inhibitors vs. Angiotensin-receptor blockers vs. their combination.

DETAILED DESCRIPTION:
Early diagnosis in children with Alport syndrome (AS) with isolated hematuria opens a "window of opportunity" for early intervention. In the Alport mouse-model, this early intervention with the ACE-inhibitor Ramipril let to a delay of kidney failure by 111%. In order to observe treatment approaches for AS in humans, this registry has been established in 2006 to collect data over several generations of Alport families across Europe. In the meantime, this registry has been expanded to "Alport XXL" via the International Alport Alliance as a global effort across all continents.

Small children with AS first develop microscopic hematuria (stage 0), proceeding to microalbuminuria (stage I), overt proteinuria (stage II), impaired kidney function (stage III) and finally can end up with kidney failure (stage IV), leading to impaired quality of life and premature death (stage V). This registry uses these stages to assess if earlier initiation of medications such as ACE-inhibition at earlier stages of disease is more effective than later therapy in delaying the time to disease progression (doubeling or tripeling of albuminuria), delaying loss of estimated glomerular filtration rate (eGFR), and if therapy improves life-expectancy.

Untreated children with autosomal-recessive AS, digenic AS, and boys with X-linked AS typically all develop kidney failure early in life. Untreated girls with X-linked AS have a 30-40% risk of kidney failure, typically later in life (40 years or older). Untreated heterozygous patients with COL4A3/COL4A4 variants typically have a less severe phenotype (in former times also called "familial benign hematuria" or "thin basement membrane nephropathy" (TBMN)) and a 1-2% risk of kidney failure.

Several interim results of this registry have been published since 2012.

Alport XXL is designed and conducted as strictly observational, non-interventional data acquisition with prospective (and in parts retrospective) data analysis. Young patients with AS in disease stages 0,I,II from all over the world are included. The renewed version from 2021 has been re-approved by the Ethics Committee of the University Medical Center Göttingen as "Alport XXL", a further development of the former European Alport Therapy Registry (AZ 10/11/06). "Alport XXL" registry and data storage are in conformity with Good Clinical Practice guidelines.

ICH-GCP-conform patient information and data exchange is secured by data transfer and cooperation agreements between all international trial centers and the coordinating principal investigator at University Medical Center Goettingen. At baseline, data collection including retrospective data is performed using a standardized, ICH-GCP-conform and pseudonymized questionnaire assessing age, sex, weight, height, mode of inheritance (X-linked, autosomal, compound heterozygous/homozygous, number of missense variants), family history, albumin in 24-hour or spontaneous urine, serum-creatinine, RAS-blockade with preparation and dose. Follow-up visits include same data than baseline plus blood-pressure, smoking-status, serum-potassium, eGFR, hearing loss and eye involvement, other symptoms such as leiomyomatosis, comorbidities and adverse events (adverse events of special interest defined as hyperkalemia, cough, hypotension, acute renal failure, malignancy, death).

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Alport syndrome (AS) by kidney biopsy or mutation analysis (or both).

Any type of genetic variant is accepted for X-linked, autosomal or digenic Alport syndrome (COL4A3, 4 or 5 genes).

Exclusion criteria:

Patients not willing to give informed consent. Patient with suspected diagnosis, whcih cannot be confirmed.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: For Alport XXL, eligible patients were children or young adults with a definitive diagnosis of AS by genetic analysis or kidney biopsy and at early stages of AS (stages 0, I or II) at baseline.
  AS stages were defined as:
  Stage 0 Microhematuria without microalbuminuria Stage I Microalbuminuria: UACR 30-300 mg/gCreatinine Stage II Proteinuria: UACR >300 with eGFR>60 ml/min/1.73m2 Stage III eGFR<60 ml/min/1.73m2 Stage IV end stage kidney failure Stage V death (from all causes)
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 1995-07; Primary Completion 2036-03-01 (Estimated); Study Completion 2036-03-01 (Estimated)

PRIMARY OUTCOMES:
age at onset of end stage kidney failure (need for renal replacement therapy) | until end of observation in 2037
  kidney disease in Alport syndrome starts at birth, age at onset of end stage kidney failure in years
life-expectancy in years (age at death) | until end of observation in 2037
  Alport syndrome starts at birth, age at death of patients in years
yearly loss of estimated glomerular filtration rate (eGFR) | until end of observation in 2037
  kidney disease in Alport syndrome starts at birth, eGFR-loss per year in ml/min/1.73m2
time in years until doubling or tripling of urinary albumin to creatinine ratio (UACR) | until end of observation in 2037
  kidney disease in Alport syndrome starts at birth; time since birth to doubling (AS stages I or II) or tripling (AS stage 0) of UACR in years.

SECONDARY OUTCOMES:
amount of albuminuria over time | until end of observation in 2037
  kidney disease in Alport syndrome starts at birth; change in albuminuria after birth
amount of proteinuria over time | until end of observation in 2037
  kidney disease in Alport syndrome starts at birth; change in proteinuria after birth
number of patients with X-chromosomal or autosomal inheritance | until end of observation in 2037
  specific genetic variant: X-linked, digenic, autosomal heterozygous, homozygous, compound heterozygous
number of patients experiencing side effects (AEs) | until end of observation in 2037
  AEs of special interest: acute kidney renal failure, angioedema, hyperkalemia, dry cough, symptomatic hypotension (orthostatic collapse) and others, and death from all causes.
number of patients with hearing loss | until end of observation in 2037
  Alport syndrome is a genetic disease, hearing loss delevops over time since birth
number of patients with eye involvement | until end of observation in 2037
  Alport syndrome is a genetic disease, eye symptoms delevop over time since birth
number of patients with positive family history of end stage kidney failure | until end of observation in 2037
  number of relatives with kidney failure
age of relatives at end stage kidney failure | until end of observation in 2037
  age of relatives at start of renal replacement therapy in years

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Gross, MD, Principal Investigator — University Hospital Goettingen
Locations (1):
- University Medical Center Göttingen, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Investigators plan to share the full data set with other researchers upon reasonable request via written cooperation agreements.

REFERENCES:
- [Background] Kashtan CE, Gross O. Clinical practice recommendations for the diagnosis and management of Alport syndrome in children, adolescents, and young adults-an update for 2020. Pediatr Nephrol. 2021 Mar;36(3):711-719. doi: 10.1007/s00467-020-04819-6. Epub 2020 Nov 6. PMID 33159213
- [Background] Weinstock BA, Feldman DL, Fornoni A, Gross O, Kashtan CE, Lagas S, Lennon R, Miner JH, Rheault MN, Simon JF; Workshop Participants. Clinical trial recommendations for potential Alport syndrome therapies. Kidney Int. 2020 Jun;97(6):1109-1116. doi: 10.1016/j.kint.2020.02.029. Epub 2020 Apr 6. PMID 32386680
- [Result] Temme J, Kramer A, Jager KJ, Lange K, Peters F, Muller GA, Kramar R, Heaf JG, Finne P, Palsson R, Reisaeter AV, Hoitsma AJ, Metcalfe W, Postorino M, Zurriaga O, Santos JP, Ravani P, Jarraya F, Verrina E, Dekker FW, Gross O. Outcomes of male patients with Alport syndrome undergoing renal replacement therapy. Clin J Am Soc Nephrol. 2012 Dec;7(12):1969-76. doi: 10.2215/CJN.02190312. Epub 2012 Sep 20. PMID 22997344
- [Result] Temme J, Peters F, Lange K, Pirson Y, Heidet L, Torra R, Grunfeld JP, Weber M, Licht C, Muller GA, Gross O. Incidence of renal failure and nephroprotection by RAAS inhibition in heterozygous carriers of X-chromosomal and autosomal recessive Alport mutations. Kidney Int. 2012 Apr;81(8):779-83. doi: 10.1038/ki.2011.452. Epub 2012 Jan 11. PMID 22237748
- [Result] Gross O, Licht C, Anders HJ, Hoppe B, Beck B, Tonshoff B, Hocker B, Wygoda S, Ehrich JH, Pape L, Konrad M, Rascher W, Dotsch J, Muller-Wiefel DE, Hoyer P; Study Group Members of the Gesellschaft fur Padiatrische Nephrologie; Knebelmann B, Pirson Y, Grunfeld JP, Niaudet P, Cochat P, Heidet L, Lebbah S, Torra R, Friede T, Lange K, Muller GA, Weber M. Early angiotensin-converting enzyme inhibition in Alport syndrome delays renal failure and improves life expectancy. Kidney Int. 2012 Mar;81(5):494-501. doi: 10.1038/ki.2011.407. Epub 2011 Dec 14. PMID 22166847
- [Result] Stock J, Kuenanz J, Glonke N, Sonntag J, Frese J, Tonshoff B, Hocker B, Hoppe B, Feldkotter M, Pape L, Lerch C, Wygoda S, Weber M, Muller GA, Gross O. Prospective study on the potential of RAAS blockade to halt renal disease in Alport syndrome patients with heterozygous mutations. Pediatr Nephrol. 2017 Jan;32(1):131-137. doi: 10.1007/s00467-016-3452-z. Epub 2016 Jul 11. PMID 27402170
- [Result] Frese J, Kettwig M, Zappel H, Hofer J, Grone HJ, Nagel M, Sunder-Plassmann G, Kain R, Neuweiler J, Gross O. Kidney Injury by Variants in the COL4A5 Gene Aggravated by Polymorphisms in Slit Diaphragm Genes Causes Focal Segmental Glomerulosclerosis. Int J Mol Sci. 2019 Jan 26;20(3):519. doi: 10.3390/ijms20030519. PMID 30691124
- [Result] Boeckhaus J, Hoefele J, Riedhammer KM, Nagel M, Beck BB, Choi M, Gollasch M, Bergmann C, Sonntag JE, Troesch V, Stock J, Gross O. Lifelong effect of therapy in young patients with the COL4A5 Alport missense variant p.(Gly624Asp): a prospective cohort study. Nephrol Dial Transplant. 2022 Nov 23;37(12):2496-2504. doi: 10.1093/ndt/gfac006. PMID 35022790
- [Result] Zhang Y, Bockhaus J, Wang F, Wang S, Rubel D, Gross O, Ding J. Genotype-phenotype correlations and nephroprotective effects of RAAS inhibition in patients with autosomal recessive Alport syndrome. Pediatr Nephrol. 2021 Sep;36(9):2719-2730. doi: 10.1007/s00467-021-05040-9. Epub 2021 Mar 27. PMID 33772369
- [Result] Boeckhaus J, Gross O. Sodium-Glucose Cotransporter-2 Inhibitors in Patients with Hereditary Podocytopathies, Alport Syndrome, and FSGS: A Case Series to Better Plan a Large-Scale Study. Cells. 2021 Jul 18;10(7):1815. doi: 10.3390/cells10071815. PMID 34359984
- [Result] Boeckhaus J, Gale DP, Simon J, Ding J, Zhang Y, Bergmann C, Turner AN, Hall M, Sayer JA, Srivastava S, Kang HG, Cerkauskaite-Kerpauskiene A, Gillion V, Claes KJ, Krueger B, de Fallois J, Walden U, Choi M, Schueler M, Mueller RU, Todorova P, Hohenstein B, Zeisberg M, Friede T, Knebelmann B, Halbritter J, Gross O. SGLT2-Inhibition in Patients With Alport Syndrome. Kidney Int Rep. 2024 Sep 24;9(12):3490-3500. doi: 10.1016/j.ekir.2024.09.014. eCollection 2024 Dec. PMID 39698346

DOCUMENTS (2):
  • Study Protocol (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT02378805/Prot_000.pdf
  • Informed Consent Form (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT02378805/ICF_001.pdf